CLINICAL TRIAL: NCT03605212
Title: Open Label, Multi-centre, Parallel Group Study to Compare the Pharmacokinetics (PK), Pharmacodynamics (PD) and Safety of Febuxostat Between Pediatric Patients (≥6<18 Years of Age) and Adults
Brief Title: Febuxostat for Tumor Lysis Syndrome Prevention in Hematological Malignancies of Paediatric Patients and Adults
Acronym: FLORET
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was stopped as per EMA waiver granted on 20July2018.
Sponsor: Menarini Group (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FLO-02; 2016-001445-61 (EudraCT Number)
Record Dates: First submitted 2018-05-29; First posted 2018-07-30 (Actual); Results first posted 2021-06-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2019-01

CONDITIONS: Tumor Lysis Syndrome
Keywords: TLS; FLO-02; Hematological Malignancies
MeSH Terms: conditions — Tumor Lysis Syndrome; Hematologic Neoplasms | interventions — Febuxostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): Febuxostat film-coated tablets 2x20 mg/QD for 7-9 days
  Interventions: Drug: Febuxostat
- Cohort 2 (Experimental): Febuxostat film-coated tablets 3x20 mg/QD for 7-9 days
  Interventions: Drug: Febuxostat
- Cohort 3 (Experimental): Febuxostat film-coated tablets 1x80 mg/QD for 7-9 days (Adenuric® 80 mg)
  Interventions: Drug: Febuxostat
- Cohort 4 (Experimental): Febuxostat film-coated tablets 1x120 mg/QD for 7-9 days (Adenuric® 120 mg)
  Interventions: Drug: Febuxostat
- Adults (Active Comparator): Febuxostat film-coated tablets 120 mg/QD for 7-9 days (Adenuric® 120 mg)
  Interventions: Drug: Febuxostat

INTERVENTIONS:
Drug: Febuxostat — Intervention is orally administered to patients in this arm.

SUMMARY:
The purpose of this study is to compare the exposure of febuxostat in pediatric patients (≥6<18 years of age) and in adults suffering from hematological malignancies at intermediate to high risk of TLS and to compare the effect in terms of serum uric acid levels.

DETAILED DESCRIPTION:
In the FLORET study it is planned to enroll 3 groups of patients in order to receive oral administration (film-coated tablets) of two different dose levels of febuxostat: children (from 6 to less than 12 years of age) will receive two different dose levels respectively; adolescents (from 12 to less than 18 years of age) will receive 80 and 120 mg/day respectively and adults (equal or major than 18 years of age) will receive 120 mg/day. The two dose levels for children and adolescents groups were to be sequentially administered, whereas the groups that will receive the first dose levels will simultaneously start the treatment at the study beginning. The individual treatment duration will be of 7 to 9 days, according to chemotherapy duration, as per Investigator's judgement.

ELIGIBILITY:
Inclusion Criteria:

male and female children of 6 to less than 12 years of age, adolescents of 12 to less than 18 years of age and adults from 18 years:

* scheduled for first cytotoxic chemotherapy cycle because of hematologic malignancies
* and at intermediate or high risk of TLS
* and with no access to rasburicase

Exclusion Criteria:

* patients with contraindications as per febuxostat summary of product characteristics
* patients with severe renal insufficiency
* patients with severe hepatic insufficiency
* patients with diagnosis of Laboratory TLS (LTLS) or Clinical TLS (CTLS)

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2018-07-25 (Actual); Study Completion 2018-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franco Locatelli, Prof, MD, Study Chair — IRCCS Ospedale Pediatrico Bambino Gesù, Piazza Sant'Onofrio, 4, 00165 Rome, IT
Locations (17):
- University Hospital Tsaritsa Yoanna, Sofia, Bulgaria
- Hungary (3):
  - Semmelweis Egyetem (paediatric), Budapest
  - Semmelweis Egyetem, Budapest
  - Debreceni Egyetem Klinikai Központ, Debrecen
- Italy (9):
  - SOC Oncologia Medica A - Centro di Riferimento Oncologico, Aviano, Pordenone
  - Policlinico S. Orsola Malpighi, Bologna
  - A.O.U.C. Azienda Ospedaliero - Universitaria Careggi, Florence
  - Azienda Ospedaliero Universitaria Meyer, Florence
  - Istituto G Gaslini Ospedale Pediatrico IRCCS, Genova
  - Azienda Ospedaliero-Universitaria Pisana, Pisa
  - IRCCS Ospedale Pediatrico Bambino Gesù, Rome
  - Ospedale Infantile Regina Margherita, Torino
  - Azienda Ospedaliera Universitaria Integrata di Verona, Verona
- Spain (4):
  - Hospital de San Pedro de Alcantara, Cáceres
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitari i Politècnic La Fe, Valencia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was screened and enrolled on 27 Feb 2017. The last patient completed the study on 16 Jul 2018. The study was conducted at 17 sites in 4 European countries.
Pre-assignment Details: A total of 31 patients was screened, of whom 30 were enrolled and 28 completed the study regularly.
  Two enrolled patients were withdrawn from study drug treatment.
Groups:
- Adults: Febuxostat film-coated tablets 1x120 mg/QD for 7-9 days (Adenuric® 120 mg)
  Febuxostat: Intervention is orally administered to patients in this arm.
Period: Baseline Period
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Adults
Started | 3 | 0 | 3 | 0 | 24
Completed | 3 | 0 | 3 | 0 | 24
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Treatment Period
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Adults
Started | 3 | 0 | 3 | 0 | 24
Completed | 2 | 0 | 3 | 0 | 23
Not Completed | 1 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: DAY 1 before first febuxostat dosing.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Adults | Total
Number analyzed (Participants) | 3 | 0 | 3 | 0 | 24 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 0 | 3 | 0 | 0 | 6
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 14 | 14
  >=65 years | 0 | 0 | 0 | 0 | 10 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.33 (1.528) |  | 14.00 (1.000) |  | 60.21 (15.376) | 50.30 (24.419)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 2 | 0 | 11 | 14
  Male | 2 | 0 | 1 | 0 | 13 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 3 | 0 | 2 | 0 | 24 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 0 | 2 | 0 | 23 | 28
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Hungary | 0 |  | 0 |  | 8 | 8
  Italy | 3 |  | 3 |  | 5 | 11
  Bulgaria | 0 |  | 0 |  | 0 | 0
  Spain | 0 |  | 0 |  | 11 | 11
Weight [Mean (Standard Deviation); unit: kg] | 26.13 (2.043) |  | 60.47 (19.747) |  | 75.60 (15.469) | 68.92 (21.369)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic (PK) Parameter: Apparent Clearance (CL/F)
Description: Apparent clearance of febuxostat from Visit 2 (Day 2) to Evaluation Visit (Visit 8, Day 8)
Time Frame: 7 days
Population: Data were not collected.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Adults
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: PK Parameter: Apparent Volume of Distribution (Vd/F)
Description: Apparent volume of distribution of febuxostat from Visit 2 (Day 2) to Evaluation Visit (Visit 8, Day 8)
Time Frame: 7 days
Population: Data were not collected.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Adults
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: PK Parameter: Absorption Rate Constant (Ka)
Description: Absorption rate constant of febuxostat from Visit 2 (Day 2) to Evaluation Visit (Visit 8, Day 8)
Time Frame: 7 days
Population: Data were not collected.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Adults
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: PK Parameter: Area Under Curve (AUC)
Description: AUC of febuxostat from Visit 2 (Day 2) to Evaluation Visit (Visit 8, Day 8)
Time Frame: 7 days
Population: Data were not collected.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Adults
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: PK Parameter: Maximum Plasma Concentration (Cmax)
Description: Maximum plasma concentration of febuxostat from Visit 2 (Day 2) to Evaluation Visit (Visit 8, Day 8)
Time Frame: 7 days
Population: Data were not collected.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Adults
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: PK Parameter: Tmax
Description: Time to Cmax from Visit 2 (Day 2) to Evaluation Visit (Visit 8, Day 8)
Time Frame: 7 days
Population: Data were not collected.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Adults
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Pharmacodynamic (PD) Parameter: Area Under the Curve of Serum Uric Acid (sUA)
Description: Area under the curve of sUA from baseline (Visit 1, Day 1) to the Evaluation Visit (Visit 8, Day 8) (AUC sUA 1-8)
Time Frame: 8 days
Population: Data were not collected.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Adults
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Assessment of Laboratory Tumor Lysis Syndrome (LTLS)
Description: Assessment of LTLS at Visit 1 (Day 1) and from Start of Chemotherapy (Visit 3, Day 3) to the Evaluation Visit (Visit 8, Day 8). LTLS is diagnosed if levels of 2 or more values of uric acid, potassium, phosphate or calcium are more than or less than normal at presentation or if they change by at least 25% from baseline.
Time Frame: 7 days
Population: Data were not collected.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Adults
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Assessment of Clinical Tumor Lysis Syndrome (CTLS)
Description: Assessment of CTLS at Visit 1 (Day 1) and from Start of Chemotherapy (Visit 3, Day 3) to the Evaluation Visit (Visit 8, Day 8). CTLS is present when LTLS is accompanied by at least one of the following significant clinical complications: increased creatinine level ≥ 1.5 upper limit of normal, cardiac arrhythmia/sudden death or seizure.
Time Frame: 7 days
Population: Data were not collected.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Adults
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Assessment of Treatment Emergent Signs and Symptoms (TESS)
Description: Assessment of incidence, severity (through Mild/Moderate/Severe scale), seriousness and treatment-causality of TESS from Screening Visit to End of Study Visit. Adverse events were assessed using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. An adverse event was considered as TESS if it occured for the first time or if it worsened in terms of seriousness or severity after first study drug intake.
Time Frame: Estimated maximum time frame: 27 days
Population: Safety population
Measure: Number; unit: Events
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Adults
Number analyzed (Participants) | 3 | 0 | 3 | 0 | 24
Events
  TESS | 50 |  | 21 |  | 70
  TESS grade >/=3 | 11 |  | 2 |  | 20
  Serious TESS | 1 |  | 0 |  | 7
  Related TESS | 4 |  | 0 |  | 0
  Related TESS grade >/=3 | 2 |  | 0 |  | 0
  Related TESS/Drug Withdrawn | 2 |  | 0 |  | 0

11. Secondary Outcome: Assessment of Participants Affected by Treatment Emergent Signs and Symptoms (TESS)
Description: Number of participants affected by TESS from Screening Visit to End of Study Visit.
Time Frame: Estimated maximum time frame: 27 days
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Adults
Number analyzed (Participants) | 3 | 0 | 3 | 0 | 24
participants | 3 |  | 3 |  | 20

12. Secondary Outcome: Performance Status (PS) Evaluation
Description: Quality of life was to be assessed by PS evaluation from Screening Visit to End of Study Visit. The Karnofsky Performance Status (KPS) scale was to be used for patients aged 16 years and older; the Lansky Play Performance Status (LPS) scale was to be used for patients aged less than 16 years. Both scales range from scores of 0 to 100 points at intervals of 10 where 0 points represent the worst outcome (KPS: 0 = death; LPS: 0 = unresponsive) and 100 points the best (KPS: 100 = normal, no complaints, no evidence of disease; LPS: 100 = fully active).
Time Frame: Estimated maximum time frame: 27 days
Population: Data were not collected.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Adults
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the entire duration of a patient's study participation, i.e. approximately 3 weeks. In addition, if after the end of the study the Investigator became aware of any AEs or follow-up in AEs already recorded, this information could be recorded in the eCRF until it was available.
Description: Adverse Events were collected during Screening, i.e. after ICF signature until DAY 1, Visit 1 before first IMP intake and specifically Treatment Emergent Signs and Symptoms (TESSs) occurring from first IMP intake at Visit 1, DAY 1 until Visit 10, DAY 14.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Adults
All-Cause Mortality (participants affected / at risk) | 1/3 | 0/0 | 0/3 | 0/0 | 0/24
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/0 | 0/3 | 0/0 | 5/24
Other Adverse Events (participants affected / at risk) | 3/3 | 0/0 | 3/3 | 0/0 | 20/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=0) | Cohort 3 (N=3) | Cohort 4 (N=0) | Adults (N=24)
Enterobacter test positiv (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Septioc shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=0) | Cohort 3 (N=3) | Cohort 4 (N=0) | Adults (N=24)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ALT increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
AST increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BP increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood triglycerides increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemoglobin decreased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell (WBC) count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 4 (4)
Language disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal rigidity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Faeces soft (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival swelling (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypo HDL cholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Data for all outcome measures were not collected due to the paucity of data in the minor patient population and in agreement with EMA with the exceptions of the secondary outcome Assessment of Treatment Emergent Signs and Symptoms (TESS).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to submitting the results of this study for publication or presentation, the Investigator will allow the sponsor at least 60 days time to review and comment upon the publication manuscript. It is agreed, that the results of the study will not be submitted for presentation, abstract, poster exhibition, or publication by the investigator until the sponsor has reviewed/commented and agreed to any publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-02): https://cdn.clinicaltrials.gov/large-docs/12/NCT03605212/Prot_SAP_000.pdf